CLINICAL TRIAL: NCT00729261
Title: A Prospective Trial of Elective Extubation in Brain Injured Patients Meeting Extubation Criteria for Ventilatory Support.
Brief Title: A Prospective Trial of Elective Extubation in Brain Injured Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Edward M. Manno M.D., Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1210-04
Record Dates: First submitted 2008-08-01; First posted 2008-08-07 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2008-08

CONDITIONS: Brain Injury
Keywords: mechanical ventilation; extubation; outcomes; brain injury
MeSH Terms: conditions — Brain Injuries | interventions — Airway Extubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- armA I (Experimental): Patients remain intubated until the patients Glasgow coma score improves to greater than 8.
  Interventions: Procedure: continued intubation
- arm 2 (Experimental): Patients that meet standard airway and ventilatory criteria for extubation but have a Glasgow coma score of less than or equal to 8 are immediately extubated.
  Interventions: Procedure: extubation

INTERVENTIONS:
Procedure: extubation — Brian injured patients that remained intubation solely because of a depressed level of consciousness were randomized into immediate extubation or delayed extubation until their level of consciousness improved.All patients met standard ventilatory, and airway criteria for extubation.
  Arms: arm 2
Procedure: continued intubation — patients remain intubated until their Glasgow coma scores improve to greater than 8.
  Arms: armA I

SUMMARY:
Identifying the optimal time of extubation in a brain injured population should improve patient outcome. Brain injured patients usually remain intubated due to concerns of airway maintenance. Current practice argues that unconscious patients need to remain intubated to protect their airways. More recent data however suggests that delaying extubation in this population increases pneumonias and worsens patient outcomes.

We designed a safety and feasibility study of randomizing brain injured patients into early or delayed extubation. The purpose was to gain insight into patient safety concerns and to obtain estimates of sample size needed for a larger study.

ELIGIBILITY:
Inclusion Criteria:

1. Resolution or improvement of any pulmonary process requiring mechanical ventilation.
2. Adequate gas exchange.
3. Adequate ventilation.
4. Respiratory rate to tidal volume ratio <105.
5. Core body temperature < 38 degrees celsius.
6. Hemoglobin > 8 grams per deciliter.
7. No sedative medications for 2 hours.

Neurological requirements included:

1. GCS ≤ 8.
2. Intracranial pressure (ICP) < 15 cm of water and a cerebral perfusion pressure (CPP) > 60 mm Hg for patients with intracranial pressure monitors.

Exclusion Criteria:

1. Age < 18 years.
2. Lack of informed consent by the patients' surrogate.
3. Dependence on mechanical ventilation for at least two weeks prior to enrollment.
4. Patients with tracheostomies.
5. Intubation instituted for therapeutic hyperventilation.
6. Planned surgical or radiological intervention within the next 72 hours.
7. Anticipated neurological or medically worsening conditions (i.e develop cerebral edema or vasospasm).
8. Patients intubated for airway preservation due to airway edema (cervical neck injuries or surgery) as opposed to airway protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-08; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Score | 6 months

SECONDARY OUTCOMES:
nosocomial pneumonias | hospital discharge
reintubations | hospital discharge
ICU length of stay | hospital discharge
hospital length of stay | hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Edward M. Manno, M.D., Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Coplin WM, Pierson DJ, Cooley KD, Newell DW, Rubenfeld GD. Implications of extubation delay in brain-injured patients meeting standard weaning criteria. Am J Respir Crit Care Med. 2000 May;161(5):1530-6. doi: 10.1164/ajrccm.161.5.9905102. PMID 10806150
- [Derived] Manno EM, Rabinstein AA, Wijdicks EF, Brown AW, Freeman WD, Lee VH, Weigand SD, Keegan MT, Brown DR, Whalen FX, Roy TK, Hubmayr RD. A prospective trial of elective extubation in brain injured patients meeting extubation criteria for ventilatory support: a feasibility study. Crit Care. 2008;12(6):R138. doi: 10.1186/cc7112. Epub 2008 Nov 10. PMID 19000302